CLINICAL TRIAL: NCT05288855
Title: A Double-Blind, Placebo-Controlled, Dose Escalation Study to Assess the Efficacy, Safety and Pharmacokinetics of Voclosporin in Adolescent and Pediatric Subjects With Lupus Nephritis
Brief Title: Voclosporin in Adolescent and Pediatric Subjects With Lupus Nephritis
Acronym: VOCAL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMB recommendation
Sponsor: Aurinia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUR-VCS-2020-03
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Adolescent Lupus Nephritis; Pediatric Lupus Nephritis
Keywords: Lupus nephritis; calcineurin inhibitors; voclosporin; adolescents; pediatrics
MeSH Terms: conditions — Lupus Nephritis | interventions — voclosporin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind (participant, care provider, investigator and outcome assessor) for period 1 and Open-label for period 2 and period 3
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Voclosporin treatment group 1 (Experimental): 2 capsules (15.8 mg) BID of voclosporin
  Interventions: Drug: Voclosporin
- Placebo treatment group 2 (Placebo Comparator): 2 capsules BID of placebo
  Interventions: Drug: Placebo Oral Capsule
- Voclosporin treatment group 3 (Experimental): 3 capsules (23.7 mg) BID of voclosporin
  Interventions: Drug: Voclosporin
- Voclosporin treatment group 4 (Experimental): Maximum dose of 2 capsules (15.8 mg) BID of voclosporin.
  Interventions: Drug: Voclosporin

INTERVENTIONS:
Drug: Voclosporin — calcineurin inhibitor
  Arms: Voclosporin treatment group 1; Voclosporin treatment group 3; Voclosporin treatment group 4
Drug: Placebo Oral Capsule — matching placebo capsule
  Arms: Placebo treatment group 2

SUMMARY:
The purpose of this study is to assess the efficacy and safety of voclosporin compared to placebo in achieving renal response following 24 weeks of therapy in adolescent and pediatric subjects with active lupus nephritis (LN).

DETAILED DESCRIPTION:
This is a 24 week, dose escalation study of voclosporin in addition to standard of care with mycophenolate mofetil (MMF) and steroids, consisting of 3 treatment periods: Period 1 is double-blind, placebo controlled receiving 15.8 mg twice daily, Period 2 is open-label receiving 23.7 mg twice daily, Period 3 is open-label receiving 15.8 mg twice daily.

ELIGIBILITY:
Key Inclusion Criteria:

* Previous diagnosis of systemic lupus erythematosus (SLE) as per the 2019 EULAR/ ACR classification criteria.
* Subjects with kidney biopsy confirmed active lupus nephritis.

Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR) <60 mL/minute/1.73 m2 at screening.
* Current or medical history of:

  * Congenital or acquired immunodeficiency.
  * Clinically significant drug or alcohol abuse prior to screening.
  * Malignant neoplasm.
  * Lymphoproliferative disease or previous total lymphoid irradiation.
  * Known severe viral infections within 3 months of screening; or known human immunodeficiency virus infection, or hepatitis B or C virus infection at any time prior to screening.
  * Active tuberculosis (TB) or known history of TB/evidence of old TB if not taking prophylaxis with isoniazid.
* Currently requiring renal dialysis (hemodialysis or peritoneal dialysis) or expected to require dialysis during the study period.
* Other known clinically significant active medical conditions, for which the condition or the treatment of the condition may affect the study assessments or outcomes.
* Currently taking or known need for any of the following medications:

  * Immunosuppression biologic agents within 12 weeks prior to randomization, cyclophosphamide, calcineurin inhibitors (CNIs) and live attenuated vaccines, initiation or dose change of ACE inhibitors/ARBs within 4 weeks prior to randomization, IV corticosteroids and IV immunoglobulin within 2 weeks prior to screening, strong CYP3A4/5 inhibitors and inducers within 2 weeks prior to randomization.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with renal response | Week 24
  Renal response defined as UPCR ≤0.5 mg/mg, eGFR ≥60 mL/min/1.73 m2 or no decrease from baseline of >20%, no rescue medication and no steroid use >10 mg/day for ≥3 consecutive days or for ≥7 days in total between week 16 to 24

SECONDARY OUTCOMES:
Time to UPCR of ≤0.5 mg/mg. | Baseline to Week 24
  Time in days to reduction in UPCR to ≤ 0.5 mg/mg
Proportion of subjects with partial renal response | Week 24
  defined as ≥50% reduction from baseline in UPCR
Time to 50% Reduction in UPCR | Baseline to Week 24
  Time in days to reduction from baseline UPCR of at least 50% Organ Class, and preferred term.
Number of treatment-emergent adverse events (TEAEs) will be summarized by treatment group | Baseline to Week 24
  Treatment-emergent adverse events will be summarized by treatment group, System Organ Class, and preferred term

CONTACTS AND LOCATIONS:
Locations (6):
- Nemours Children's Hospital, Orlando, Orlando, Florida, United States
- Clinica de la Costa S.A.S, Barranquilla, Atlántico, Colombia
- Yokohama City University Hospital, Yokohama, Kanagawa, Japan
- Mexico (2):
  - Centro de Especialidades Medicas del Sureste, Mérida, Yucatán
  - Hospital Infantil de México Federico Gómez, Mexico City
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No